CLINICAL TRIAL: NCT05471765
Title: Effects of Continuous Positive Airway Pressure Therapy Withdrawal in Patients With Obstructive Sleep Apnea: A Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Siraj Omar Wali, Director of Sleep Medicine and Research Center, Professor of Medicine, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 241-20
Record Dates: First submitted 2022-06-29; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate Obstructive Sleep Apnea (Experimental): Patients whom have an apnea/hypopnea index above fifteen are classified to have moderate obstructive sleep apnea
  Interventions: Device: Withdrawal of Continuous Positive Airway Pressure device; Device: Alternation usage of Continuous Positive Airway Pressure Device
- Severe Obstructive Sleep Apnea (Experimental): Patients whom have an apnea/hypopnea index with a result higher than thirty are considered to have severe obstructive sleep apnea
  Interventions: Device: Withdrawal of Continuous Positive Airway Pressure device; Device: Alternation usage of Continuous Positive Airway Pressure Device

INTERVENTIONS:
Device: Withdrawal of Continuous Positive Airway Pressure device — After completing one month of therapeutic management with The Continuous Positive Airway Pressure device and have controlled OSA defined as Apnea Hypopnea Index (AHI) of < 5 while on treatment. At random, a group of participants will cease to use the Continuous Positive Airway Pressure. And they'll have weakly clinic visits where they will fill the Epworth Sleepiness Scale, check their blood pressure, heart rate and undergo Polysomnography for 4 weeks.
Device: Alternation usage of Continuous Positive Airway Pressure Device — After completing one month of therapeutic management with The Continuous Positive Airway Pressure device and have controlled OSA defined as Apnea Hypopnea Index (AHI) of < 5 while on treatment. Randomly, these patients will alternatively use The Continuous Positive Airway Pressure device every other day (e.g. They will use the device 4 days and not use it for 3 days of the week) and they'll have weakly clinic visits where they will fill the Epworth Sleepiness Scale, check their blood pressure, heart rate and undergo Polysomnography for 4 weeks.

SUMMARY:
Study design (e.g., double-blind:

A randomized, open-labeled, controlled, parallel-group study.

Sixty patients will be recruited with moderate to severe Obstructive Sleep Apnea (OSA), previously adherent to CPAP therapy and have controlled OSA defined as Apnea Hypopnea Index (AHI) of < 5 while on treatment. Patients will be divided into two groups after completion of Therapeutic CPAP, Who will continue on same CPAP therapy for 4 weeks they will be randomized into two groups:

1. NO CPAP (NOCPAP Group): Who will stop using the CPAP device.
2. Intermittent CPAP (Int-CPAP Group): Who will use the CPAP device every other night.

This trial will also evaluate the effects of CPAP withdrawal (complete or partial) on excessive day time sleepiness (EDS), apnea hypopnea index (AHI), Heart Rate and Blood Pressure.

DETAILED DESCRIPTION:
Obstructive sleep apnea syndrome (OSAS) is a common sleep-related breathing disorder, which is characterized by transient interruption of ventilation during sleep caused by complete or partial collapse of the upper airway. Many risk factors are identified such as: male gender, large neck circumference, smoking, excessive alcohol intake and high Body Mass Index (BMI).

The prevalence of OSAS in Saudi Arabia is about 4% and 1.8% in males and females, respectively, and it is associated with many comorbidities like type 2 DM, ischemic heart disease, congestive heart failure, hypertension and depression.

Continuous positive airway pressure (CPAP) is considered the gold standard treatment for moderate to severe (OSA) as it works as a pneumatic splint of the collapsible airway and it may induce anatomical and functional changes of the upper air way muscles. Treatment with CPAP was reported to decrease daytime sleepiness, and improve the quality of life among sleep apnea patients. However, its impact on other outcomes such as hypertension was modest but clinically significant and it may has no impact on other major cardiovascular outcomes such as cardiovascular mortality, acute coronary syndrome, stroke, transient ischemic attack or hospitalization for heart failure even in patients with established coronary artery disease, and the same result was seen in two recently published meta-analyses.

The widely used definition of acceptable adherence to the CPAP is 4 hours per night for more than 70% of all monitored days or 5 days per week. However, this definition was based on experts' opinion and the knowledge about human sleep. Many studies showed that the 4 hours cut-off was the minimum required amount of time to gain significant improvement from CPAP use and there was a linear dose response relationship with greater benefit observed with increasing nightly use.

However, few studies conducted to assess the effect of CPAP withdrawal following long term treatment of OSAS with conflicting results. The residual effects of CPAP after withdrawal has been controversial in the medical literature. Although some studies suggest that there is some form of reversibility associated with CPAP compliance which leads to improvement in subjective and objective assessment of sleepiness, however, other reports revealed that CPAP withdrawal is associated with a rapid recurrence of OSAS. Rossi et al reported that in 71% of the study population, CPAP withdrawal for four nights was associated with relapse of OSA. However, 10 % remained in remission after 2 weeks of treatment withdrawal. Moreover, we could not find a study that evaluated an intermittent CPAP therapy after a long period of adherence. However, Issa & Sullivan reported that after 2-3 month of daily CPAP use, patients who use CPAP on intermittent 3-4 nights "on" and 2-3 nights "off were able to maintain good day time function, which maybe a reflection of a less fragmented sleep, thus an adequately controlled OSAS.

Nevertheless, the withdrawal of CPAP raises an ethical concern. However, several reports support the relieve from this fear. Studies of Short-term CPAP withdrawal revealed that it was not associated with any impairment of coronary endothelial function, or raise of stress hormones and markers of vascular inflammation. In addition, the recent Australian and the SAVE studies that were quoted before revealed no significant effect of CPAP on preventing secondary cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 75 years, AHI > 15 based on PSG An Epworth Sleepiness Scale (ESS) of >10, (At base line before treatment ) Stable BMI: defines as BMI that has been stable with no more than 10 % changes. Currently on CPAP therapy for more than or equal of 6 months Compliance with CPAP defined as more than 4 hours per night for an average of 5 nights per week or ≥ 70% of all recorded days Current ESS score of <10.

Exclusion Criteria:

* Patients with ventilatory failure, Cheyne-Stokes breathing, unstable and untreated coronary or peripheral artery disease, severe and inadequately controlled arterial hypertension, or a history of any sleep-related accident, or who were current professional drivers, were excluded from the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Achieving a desaturation SPO2 index of >10 or AHI of >5 | six months
  Achieving a desaturation SPO2 index of >10 or AHI of >5

SECONDARY OUTCOMES:
Recurrence of excessive sleepiness daytime symptoms | six months
  * lack of concentration
  * inability to retain new information
  * dozing off or feeling sleepy while driving, sitting or talking
  * fogy mind
  * feeling sleepy despite long hours of sleeping

OTHER OUTCOMES:
Primary safety endpoint (study stopping rules): The study will be discontinued for any participants if any of the following developed | six months
  Symptoms of Obstructive Sleep Apnea Excessive daytime sleepiness Recurrent awakening from sleep Drop in oxygen saturation during sleep that will be measured every 4 nights. Documented AHI of more than 5 in the repeated PSG If the patient developed any acute sickness that required medical attention

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wali SO, Batawi G, Kanbr O, Butt NS, Yasawy MA, Alqaidi D, Alhejaili F, Alshumrani R, Gozal D. Impact of continuous positive airway pressure therapy withdrawal in patients with obstructive sleep apnea: a randomized controlled trial. Sleep Breath. 2025 Apr 1;29(2):146. doi: 10.1007/s11325-025-03309-z. PMID 40167853